CLINICAL TRIAL: NCT00411788
Title: A Phase II Study of Rapamycin (Rapamune, Sirolimus) and Trastuzumab (Herceptin) for Patients With HER-2 Receptor Positive Metastatic Breast Cancer
Brief Title: A Phase II Study of Rapamycin and Trastuzumab for Patients With HER-2 Receptor Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0605001396
Record Dates: First submitted 2006-12-14; First posted 2006-12-15 (Estimated); Results first posted 2016-09-21 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
Keywords: HER-2 positive; breast cancer; HER-2 positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Sirolimus; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sirolimus and trastuzumab (Experimental): Patients received oral sirolimus 6 mg daily in combination with weekly trastuzumab administered intravenously with a loading dose of 4 mg/kg followed by 2 mg/kg weekly in a 28-day cycle. A subsequent amendment allowed trastuzumab to be administered every 3 weeks for patient convenience, with a loading dose of 8 mg/kg followed by a 6 mg/kg in a 21-day cycle. Sirolimus was administered at a 6 mg oral daily dose. Cycles were repeated on an every 21 or 28-day schedule until disease progression, unacceptable toxicity, or the development of any of the criteria for study removal. Doses were reduced or discontinued based on tolerability.
  Interventions: Drug: Rapamycin; Drug: Trastuzumab

INTERVENTIONS:
Drug: Rapamycin — oral rapamycin 6 mg daily
  Other Names: Rapamune; Sirolimus
Drug: Trastuzumab — Trastuzumab 4 mg/kg will be administered (intravenous) on day 1, and this will be followed by weekly dose of 2 mg/kg starting day 8.
  Other Names: Herceptin

SUMMARY:
Rapamune (generic name: Sirolimus®) is a drug that has been approved by the Food and Drug Administration (government) for use in patients receiving a kidney transplant to prevent the patient's body from rejecting the transplanted kidney. It has shown antitumor effects in the laboratory, but has not been approved at this time for the treatment of cancer. Herceptin is a new form of chemotherapy that has been approved by the Food and Drug Administration for the treatment of breast cancer.

This study is designed to evaluate the effect and safety of combining Rapamune and Herceptin on breast cancer. Rapamune and Herceptin are being combined because results from our laboratory studies suggest that the combination of the two drugs is superior to either drug used alone. Results from laboratory studies performed at other institutions suggest that adding Rapamune to Herceptin may also reverse the resistance to Herceptin. Although there has been extensive experience using Herceptin alone and Rapamune alone in human subjects, the combination of Herceptin and Rapamune has not been previously evaluated. In addition, we hope to better understand how these treatments work against an individual woman's tumor by analyzing tissue samples before, and during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed HER2 overexpressing (IHC 3+ and/or FISH +) metastatic breast cancer with measurable disease. Patients with either HER2 3+ positive tumors by immunohistochemistry (Dako Herceptest®) or gene amplification (> 2 copies) by fluorescence in-situ hybridation (FISH) are eligible.
* Progression following at least 8 weeks of standard doses of Herceptin or a Herceptin containing regimen.
* Off Herceptin for a minimum of 2 weeks.
* Patients must have measurable disease as defined by RECIST guidelines (the lesion that will be biopsied on study cannot be the only measurable lesion).
* Life expectancy > 3 months
* Age ≥18 years
* ECOG performance status ≤2
* Adequate bone marrow function as indicated by the following:

  * ANC ≥1500/µL
  * Platelets ≥100,000/µL
  * Hemoglobin ≥9 g/dL
* Adequate liver function, as indicated by bilirubin ≤1.5 x ULN, AST or ALT <2x ULN.
* Adequate renal function, as indicated by creatinine <1.5 x upper limit of normal (ULN)
* Ability to understand and the willingness to sign a written informed consent.
* Adequate birth control: Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and must have a negative serum or urine pregnancy test within 1 week prior to beginning treatment on this trial. Pregnant and nursing patients are excluded because the effects of the combination of Rapamycin on a fetus or nursing child are unknown. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Fasting serum cholesterol <350 mg/d L and triglycerides < 400 mg/ d L.
* Biopsy is required but patients or physicians may opt out of this part of the trial if sufficient justification is provided. Justification must be provided to the PI in writing indicating excessive physical risk or psychological trauma if biopsy is undertaken.

Exclusion Criteria:

* Active infection or treatment for systemic infections within 14 days of enrollment
* Patients with active brain metastases requiring treatment, inclusive but not limited to surgery, radiation, and corticosteroids (patients with asymptomatic non- progressing brain metastasis who have completed treatment ≥30 days before enrollment and without evidence of progression on a post treatment MRI may be considered for the study).
* Pregnant or lactating women
* Prior chemotherapy within the last 4 weeks (last 6 weeks for nitrosureas/mitomycin)
* Prior radiation therapy within the last 4 weeks; prior radiation therapy to indicator lesion (unless objective disease recurrence or progression within the radiation portal has been documented since completion of radiation).
* Prior therapy with rapamycin, rapamycin analogs, or experimental agents targeting mTOR.
* Concomitant malignancies or previous malignancies within the last 5 years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* Ejection fraction <50% or below the lower limit of the institutional normal range, whichever is lower
* Hypersensitivity to trial medications
* Patients may not be receiving any other investigational agents within 30 days before enrollment.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because the investigational agents may have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued if the mother is treated.
* HIV-positive patients are ineligible because these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy and the potential pharmacokinetic interaction between antiretroviral therapy and the investigational agents.
* Use of all herbal and alternative medications within 4 weeks. All herbal and alternative medications should be discontinued while on study, these include but not limited to: Hydrastis canadensis (goldenseal) - Uncaria tomentosa (cat's claw) - Echinacea angustifolia roots - trifolium pratense (wild cherry) - matricaria chamomila (chamomile) - Glycyrrhiza glabra (licorice) - dillapiol - naringenim.
* Use of any of these medications within 4 weeks; cyclosporine, diltiazen, ketoconazole, rifampin, fluconazole, delavirdine, nicardipine, pioglitazone, and sulfonamides, erythromycin, clarithromycin, itraconazole, erythromycin, metoclopramide, nevirapine, phenobarbital, phenytoin, indinavir, fosamprenavir, nefazadone, St Johns Wort.
* Consumption of grapefruit juice is prohibited during the study.
* Use of warfarin (Coumadin), immunosuppressive agents or chronic oral, intravenous or topical steroid

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maysa Abu-Khalaf, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Yale Comprehensive Cancer Center at Yale University School of Medicine, New Haven, Connecticut

RESULTS

PARTICIPANT FLOW:
Groups:
- Rapamycin and Trastuzumab: Patients received oral rapamycin/sirolimus 6 mg daily in combination with weekly trastuzumab administered intravenously with a loading dose of 4 mg/kg followed by 2 mg/kg weekly in a 28-day cycle. A subsequent amendment allowed trastuzumab to be administered every 3 weeks for patient convenience, with a loading dose of 8 mg/kg followed by a 6 mg/kg in a 21-day cycle. Sirolimus was administered at a 6 mg oral daily dose. Cycles were repeated on an every 21 or 28-day schedule until disease progression, unacceptable toxicity, or the development of any of the criteria for study removal. Doses were reduced or discontinued based on tolerability.
Period: Overall Study
Arm/Group | Rapamycin and Trastuzumab
Started | 11
Completed | 9
Not Completed | 2
Not completed — Protocol Violation | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Eleven patients were enrolled from study start date until February 2010.
Arm/Group | Rapamycin and Trastuzumab
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 57 [38 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Are Progression-free (CR, PR and Stable Disease)
Description: To determine the clinical activity of oral daily rapamycin administered in combination with weekly intravenous trastuzumab in patients with HER2 overexpressing advanced breast cancer, the primary outcome is to determine the proportion of patients who are progression-free at 16 weeks, defined by complete response (CR), partial response (PR), or stable disease (SD).who are progression free at 16 weeks, defined by complete response (CR), partial response (PR), or stable disease (SD). Response objectives assessed using response evaluation criteria (RECIST) 1.0
  This primary outcome was reworded from its original format when results were entered.
Time Frame: 16 weeks
Population: Nine patients were evaluable for response assessment. Two patients withdrew from study before first response assessment (one for noncompliance and the other for toxicity).
Measure: Number; unit: participants
Arm/Group | Sirolimus and Trastuzumab
Number analyzed (Participants) | 9
participants | 4

2. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was determined according to RECIST criteria, duration of response, and time to progression in patients with HER2 overexpressing advanced breast cancer receiving trastuzumab and rapamycin. The objective response rate (ORR) by response evaluation criteria (RECIST) 1.0, duration of response, safety, and pharmacodynamic endpoints.
  This secondary outcome measure was reworded from its original submission when results were entered.
Time Frame: study completion up to 58 weeks
Measure: Number; unit: participants
Arm/Group | Sirolimus and Trastuzumab
Number analyzed (Participants) | 9
participants | 1

3. Secondary Outcome: Incidence of Cardiac Dysfunction
Description: This safety measure was used to determine the number of patients treated with the combination of trastuzumab and rapamycin with cardiac dysfunction.
  This secondary outcome measure was reworded from its original version when results were entered.
Time Frame: study completion up to 58 weeks
Population: Safety population consisting of 9 of 11 patients that received treatment following first dose.
Measure: Number; unit: participants
Arm/Group | Sirolimus and Trastuzumab
Number analyzed (Participants) | 9
participants | 1

4. Secondary Outcome: To Determine Pre and Post Therapy Changes in the Levels, Phosphorylation Status and/or Subcellular Localization of the Affected Signal Transduction Molecules HER2, Akt, S6K and 4EBP1 in Blood and Tumor Tissues
Description: These data were not collected and analyzed as described here in the initial protocol submission.
Time Frame: Upon completion of study
Arm/Group | Sirolimus and Trastuzumab
Number analyzed (Participants) | 0

5. Secondary Outcome: To Determine if Currently Available RNA Expression Profiles Associated With Response to Herceptin Will be Predictably Altered in Tumors Treated With Trastuzumab and Rapamycin, and Will Further Elucidate the Mechanism of Synergy of These Two Agents
Time Frame: study completion
Population: This outcome measure was not collected nor analyzed due to study closure and low sample size.
Arm/Group | Sirolimus and Trastuzumab
Number analyzed (Participants) | 0

6. Secondary Outcome: To Evaluate the Use of FDG-PET as an Early Predictor of Response to the Combination of Rapamycin and Trastuzumab, be Assessing Changes in Glucose Metabolism and Cell Viability Between Pre- and Post-treatment
Time Frame: Upon completion of study
Population: This outcome measure was not collected nor analyzed due to study closure and low sample size.
Arm/Group | Sirolimus and Trastuzumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected in aggregate through the end of the study (up to 58 weeks).
Arm/Group | Sirolimus and Trastuzumab
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus and Trastuzumab (N=9)
Hyperglycemia (Endocrine disorders) | 1 (1)
Cardiac Dysfunction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus and Trastuzumab (N=9)
Leukopenia (Blood and lymphatic system disorders) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 8 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)
Nail Changes (Skin and subcutaneous tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Mucositis (Infections and infestations) | 5 (5)
Xerostomia (General disorders) | 1 (1)
Dysgeusia (General disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridemia (Blood and lymphatic system disorders) | 2 (2)
Hyperglycemia (Endocrine disorders) | 2 (2)
AST/ALT (Endocrine disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes